CLINICAL TRIAL: NCT00597311
Title: Preoperative Chemoradiation Versus Short Term Radiation Alone With Delayed Surgery for Stage II and III Resectable Rectal Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaunas University of Medicine (Other)
Responsible Party: Tadas Latkauskas, Kaunas University of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BE-2-48; 137/2006
Record Dates: First submitted 2008-01-09; First posted 2008-01-18 (Estimated); Last update posted 2008-01-18 (Estimated); Status verified 2008-01

CONDITIONS: Primary Rectal Cancer
Keywords: rectal cancer; radiotherapy; radiochemotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): preoperative short term radiation group 5x5 Gy and surgery after 6 weeks
  Interventions: Radiation: radiotherapy
- 2 (Experimental): preoperative chemoradiotherapy group 50Gy + 5FU/Lv and surgery after 6 weeks.
  Interventions: Radiation: radiotherapy

INTERVENTIONS:
Radiation: radiotherapy — 1. Short term radiotherapy 5x5 Gy during 5 days
  2. Chemoradiotherapy 50 Gy + 5Fu/Lv

SUMMARY:
Trial compares two preoperative stage II and III rectal cancer treatment strategies: short term radiotherapy 5x5 Gy and delayed surgery after 6 weeks versus conventional chemoradiotherapy 50 Gy + 5Fu/Lv and surgery also after 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed stage II and III rectal cancer less than 15 cm from anal verge
* less than 80 years old
* no other cancer during 5 years period
* compensate cardiovascular, pulmonary, hepatic and renal functions.

Exclusion Criteria:

* stage I or IV rectal cancer
* other cancer in 5 years period
* radiotherapy or chemotherapy in anamnesis
* not compensate cardiovascular, pulmonary, hepatic or renal functions, neurological, psychiatric disease, sepsis, etc.
* pregnancy or baby feeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2007-01; Primary Completion 2012-01 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
5 years overall and disease free survival | 5 years
recurrence rate | 5 years

SECONDARY OUTCOMES:
pathological "complete response" and downstaging rates | 5 years
Impact on sphincter sparing operation rates | 5 years
morbidity and mortality rates | 5 years
Impact on quality of surgical resection | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Dainius Pavalkis, professor, Principal Investigator — Kaunas Medical University
Locations (1):
- KMUH, surgery department, Kaunas, Lithuania

REFERENCES:
- [Derived] Latkauskas T, Pauzas H, Kairevice L, Petrauskas A, Saladzinskas Z, Janciauskiene R, Gudaityte J, Lizdenis P, Svagzdys S, Tamelis A, Pavalkis D. Preoperative conventional chemoradiotherapy versus short-course radiotherapy with delayed surgery for rectal cancer: results of a randomized controlled trial. BMC Cancer. 2016 Dec 1;16(1):927. doi: 10.1186/s12885-016-2959-9. PMID 27903247